CLINICAL TRIAL: NCT00434239
Title: A Pilot Study of the Combination of Lenalidomide (Revlimid®) With Two Different Dose Levels of Short Term Administration of Recombinant Human Stem Cell Factor (rhSCF; Ancestim) for Myelodysplasia.
Brief Title: Lenalidomide and Recombinant Human Stem Cell Factor for Treatment of Myelodysplasia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06/49
Record Dates: First submitted 2007-02-11; First posted 2007-02-13 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Myelodysplasia
Keywords: Myelodysplasia; Lenalidomide; Ancestim; Pilot trial; Biomarkers
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts | interventions — Lenalidomide; ancestim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment: Lenalidomide and Ancestim (Experimental): Drug: Lenalidomide + Ancestim Dose level 1. Lenalidomide 10mg orally daily days 1-21/ 28 day cycle Ancestim 10mc/kg subcutaneously daily for 7 days for cycle 3 only 10mg orally daily days 1-21/ 28 day cycle. Dose level 2 Ancestim 20mc/kg subcutaneously daily for 7 days for cycle 3 only 10mg orally daily days 1-21/ 28 day cycle
  Interventions: Drug: Lenalidomide + Ancestim

INTERVENTIONS:
Drug: Lenalidomide + Ancestim — Dose level 1. Lenalidomide 10mg orally daily days 1-21/ 28 day cycle Ancestim 10mc/kg subcutaneously daily for 7 days for cycle 3 only 10mg orally daily days 1-21/ 28 day cycle. Dose level 2 Ancestim 20mc/kg subcutaneously daily for 7 days for cycle 3 only 10mg orally daily days 1-21/ 28 day cycle
  Other Names: Revlimid; rhSCF

SUMMARY:
This study is mainly assessing the safety of Revlimid in combination with Ancestim (recombinant human stem cell factor) in patients with symptomatic myelodysplasia. Of those two compounds, Revlimid has been shown to be an active drug in myelodysplasia. Clinical responses will also be assessed.

DETAILED DESCRIPTION:
Aim: The primary objective is to assess the safety of Revlimid in combination with Ancestim in patients with symptomatic myelodysplasia. The secondary objectives are: Duration of response and assessment of changes in gene expression profile of bone marrow samples from patients undergoing such treatment.

Potential Significance: Myelodysplastic syndromes (MDS) are malignant hematopoietic stem cell disorders. Prognosis can be estimated by use of the International Prognostic Scoring System (IPSS) which divides patients into low, intermediate-1, intermediate-2, and high-risk groups with corresponding median survival times of 5.7 years, 3.5 years, 1.2 years, and 0.4 years, respectively. There is currently no standard treatment for MDS and management is often purely symptomatic with transfusion of blood products and antibiotic treatment of infections.

A recent phase II study however has shown significant response rates with Revlimid as a single agent in patients with MDS. The total response rate was 56%. The effects of Revlimid and SCF on hematopoietic progenitors cells were examined in vitro. RhSCF and Revlimid were shown to be synergistic in stimulating the proliferation of hematopoietic progenitor cells and their precursors in vitro, thereby forming the rationale for this study.

Research Plan: This is a single-centre, open label, single-arm, non-comparative study, in which 25 patients will be enrolled. The study will include patients who meet all the inclusion and none of the exclusion criteria, as per the respective protocol section.

The patients will be enrolled sequentially to receive 2 different dose levels of Ancestim with a fixed dose of Revlimid. This will determine the feasibility and tolerability of the combination of Revlimid and Ancestim. Patients will start with an 8 week course of single agent Revlimid as 10mg daily oral treatment day 1-21 in a 28 day cycle. If patients do not achieve a complete remission on single agent Revlimid they will start on Ancestim s.c. injections. Two dose levels of Ancestim (10 and 20 mcg/kg s.c. daily for 7 days) will be evaluated.

Safety: Safety will be assessed by the reporting of adverse events (starting with the first study-related procedure, during treatment, and for a period of 60 days following discontinuation of treatment). The intensity of the adverse events will be assessed using National Cancer Institute common toxicity criteria. All adverse events will be recorded on the case report forms (CRFs). Furthermore, assessments of physical (including neurological / peripheral neurological) examinations, vital signs measurements, and haematology and clinical chemistry tests will be used to monitor safety. Clinically relevant changes in laboratory safety tests, vital signs, and physical examinations will be recorded as adverse events. The adverse event sections of the CRFs will be submitted to a representative of the sponsor at the end of each treatment cycle. Serious adverse events will be reported as they occur, on forms provided by the sponsor.

Efficacy: Response to treatment will be assessed according to the guidelines of the international working group to standardize response criteria for myelodysplastic syndromes. This will be done on bone marrow biopsies (including cytogenetic analyses) and peripheral blood counts. An additional scientific investigation will examine gene-expression profiles of bone-marrow and blood samples at different time points and will try to correlate those with response to treatment. Concomitant in-vitro studies will assess surrogate markers of response.

Statistical Methods: Adverse events, serious adverse events, transfusion requirements, response data and Karnofsky performance status data will be summarized.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age >18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Patients must have a confirmed myelodysplastic syndrome regardless of subgroup according to the WHO classification and their prognostic group. Patients with treatment associated MDS are allowed on this study, however the number is restricted to 10 (50% of patients anticipated to receive combination treatment). Patients with CMML are eligible but restricted in number to up to 3 in total.
5. The patients must have either:

   1. symptomatic anemia as defined as Hb < 10g/dl OR
   2. transfusion-dependent anaemia as defined as requiring more than 4 units of packed red blood cells over 8 weeks
6. All previous cancer therapy, including erythropoietin, thalidomide and other experimental therapies must have been discontinued at least 4 weeks prior to treatment in this study.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or lactating females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide.
6. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
7. Any prior use of Revlimid or SCF.
8. Concurrent use of other anti-cancer agents or treatments including erythropoietin.
9. Known positive for HIV or infectious hepatitis, type B or C.
10. Mast cell diseases (systemic mastocytosis, urticaria pigmentosa or diffuse cutaneous mastocytosis)
11. History of severe anaphylaxis, asthma, recurrent urticaria, recurrent angiooedema
12. Known hypersensitivity against to Escherichia coli derived products.
13. Prior chemotherapy or stem cell transplantation for the treatment of myelodysplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2011-05 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Toxicity as defined by NCI-CTCv3.0 | 3 years

SECONDARY OUTCOMES:
Response | 3 years
Pharmacodynamics | defined in protocol
Change in Biomarkers | defined in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Miles Prince, Prof., Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia